CLINICAL TRIAL: NCT04304014
Title: Assessment of the Impact of Type of Probiotic, Delivery Type and Feeding Type on Baby's Microbiota After Dysbiotic Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Óscar García-Algar, Principal Investigator, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro-Care 3
Record Dates: First submitted 2020-03-04; First posted 2020-03-11 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Dysbiosis
Keywords: probiotic; microbiota; newborn
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both probiotic products will be provided in their commercial form. Both products will be individually placed inside opaque bags so that the investigator can not recognize the external case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri (Experimental): Group that will receive L. reuteri one dose per day in an oral suspension
  Intervention: Dietary Supplement: L. reuteri
  Interventions: Dietary Supplement: L. reuteri
- B. longum and P. Pentosaceus (Experimental): Group that will receive B. longum and P. Pentosaceus one dose per day in an oral suspension.
  Intervention: Dietary Supplement: B. longum and P. Pentosaceus

INTERVENTIONS:
Dietary Supplement: L. reuteri — (10^8 CFU) once a day
  Arms: L. reuteri
Dietary Supplement: B. longum and P. Pentosaceus — (10^9 CFU) once a day

SUMMARY:
This study aims to determine the effect of three factors (delivery type, feeding type and the use of two different dietary supplements) on rebiosis after disbiotic delivery. This is a randomized, single-blinded study with two parallel arms. Group 1 will receive L. reuteri (10^8 CFU) once a day, group 2 will receive B. longum and P. Pentosaceus (10^9 CFU) once a day.

DETAILED DESCRIPTION:
Gut colonization during the first days of life represents the start of the infant's own microbiota. This process is influenced by different factors: delivery type, feeding type, antibiotic treatment, etc. On the one hand, vaginally delivered babies are in contact with mother's vaginal and faecal microbiota. This fact will drive a neonatal gut colonization composed of vagina-associated bacteria. In contrast, babies born by C-section are more susceptible to be colonized by microorganisms present in the mother's skin. On the other hand, antibiotic administration during vaginal delivery also produces alterations in the vaginal microbiota of the mother. Described scenarios have been correlated to immunological and metabolic diseases such as asthma, allergies, diabetes or obesity. Moreover, disbiosis has also been associated to functional gastrointestinal disorders (FGID) in babies such as infant colic and functional constipation. After a disbiotic delivery, medical doctors usually recommend the use of probiotics to prevent rebiosis. Since the probiotics.

L. reuteri, and B. longum and P. Pentosaceus have shown efficacy on FGID amelioration in previously published articles, these two probiotics were selected for the present study. All together, this study aims to characterize the role of three different parameters: type of probiotic, delivery type and feeding type.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants up to 25 days of life
* Infants with adequate weight according to the gestational age.
* Infants born by vaginal delivery whose mother was given antimicrobial prophylaxis or infants born by C-section.
* Gestational birth equal or greater than 37 weeks.
* Exclusive or almost exclusive breastfeeding (understanding almost exclusive the one in which there is a maximum of one formula feeding per day) or mixed feeding (in which there is more than one formula feeding per day).

Exclusion Criteria:

* Infants with smoker mother during pregnancy and after delivery.
* Infants whose parents cannot follow the study requirements
* Infants who have suffered neonatal admission or have suffered or suffer necrotizing enterocolitis, infectious disease, congenital malformation, short bowel syndrome or any serious illness.
* Infants who have taken probiotics before the start of the trial or who take formula with probiotics.
* Breast-fed infants whose mothers have taken probiotics within the two weeks before study inclusion.
* Infants who ingest special formulas as extensively hydrolysed formulas.
* Breast-fed infants whose mothers have excluded dairy products and egg products in their diet during breastfeeding
* Infants who take specific medication for the treatment of functional digestive disorders: antacids (type IBP or H2 blockers), laxatives (PEG, lactulose, magnesia), lactase and simethicone at the time of inclusion.
* Infants undergoing therapies with acupuncture, homeopathy, medicinal herbs, anti-inflammatories and antispasmodics at the time of inclusion.

Max Age: 25 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Relative abundance of bifidobacteria | 1 month
  Changes in the relative abundance of bifidobacteria in stool microbiota after 1 month of supplementation, measured with metagenomic techniques.

SECONDARY OUTCOMES:
Number of regurgitations by questionnaire included in patients' diary | 3 months
  Number of regurgitations will be documented by the parents each week for 3 months in patients diary
Number of constipation episodes by questionnaire included in patients' diary | 3 months
  Number of constipation episodes will be documented by the parents each week for 3 months in patients' diary
Number of infant colic episodes by questionnaire included in patients' diary | 3 months
  Number of constipation episodes will be documented by the parents each week for 3 months in patient's diary
Metagenomic analysis of total gut microbiota | 1 month
  This measure includes all bacteria detected in feaces by metagenomic analysis. Faecal samples will be collected at baseline and 1 month after probiotic treatment. Analysis will comprise changes in the relative abundance of B. longum and P. Pentosaceous as well as the order Bifidobacteriales, Lactobacillales , Bacteroidales and Enterobacterales. In addition, the proportion (Bifidobacteriales + Lactobacillales + Bacteroidales) will be determined
Respiratory, gastrointestinal infections and use of medication by questionnaire included in patients' diary | 3 months
  Number of respiratory, gastrointestinal infections and use of medication episodes will be documented by the parents each week for 3 months in patient's diary
Anxiety and depression by the validated Hospital Anxiety and Depression scale (HADS) | 3 months
  Anxiety and depression levels of the father and mother will be evaluated at baseline and 3 months after probiotic treatment through the Hospital Anxiety and Depression Scale (HADS) questionnaire will be.
  Odd questions (assess anxiety). Even questions (assess depression). Score less than or equal to 7 = no case. 8-10 = doubtful case Score equal to or greater than 11 = case
Extra visits to paediatrician/emergency by questionnaire included in the patient's diary | 3 months
  Number of paediatric visits and / or emergency access will be documented each week in the patient's diary during the 3 months of treatment
Number of Participants With Treatment-Related Adverse Events | 3 months
  Adverse events will be documented weekly in the patient's diary during the 3 months of treatment.
Levels of IgA in faeces | 1 month
  changes in IgA in faeces from baseline to 1 month of treatment
Weight evolution by the paedatrician in study visits | 3 months
  Changes on baby's body weight from baseline to 3 months of probiotic treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Fundación HM Hospitales (Hospital HM Puerta Sur), Madrid, Madrid
  - Neonatal Unit, Hospital Clinic-Maternitat, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided